CLINICAL TRIAL: NCT05277324
Title: The Effect of Wearing Facial Masks on Skin Parameters During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Dario Leskur, Assistant professor, University of Split, School of Medicine
Other Study IDs: 2181-198-03-04-22-0010
Record Dates: First submitted 2022-03-10; First posted 2022-03-14 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Skin Condition; Skin Inflammation; Facial Skin Changes
MeSH Terms: conditions — Skin Diseases; Dermatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Protective facial mask — Participants, students of health related professions, who wear protective facial mask daily during their internship/practice in health institutions.

SUMMARY:
The global coronavirus disease pandemic (COVID-19) has led to an increased need to wear protective equipment such as wearing face masks and practicing hygiene measures such as more frequent use of antiseptics. These measures can lead to changes in the skin, the development of new inflammatory skin diseases or exacerbation of existing ones, with health professionals especially under the risk of developing these changes. Changes in facial skin due to wearing masks have been observed in a number of studies, however, part of the study was based solely on subjects' self-assessment or clinical assessment, and only a small part on objective measurements of skin parameters. Also, the impact of prolonged masks' use have not been investigated.

The aim of these study was to investigate the effects of constant, long-term use of protective masks on facial skin.

ELIGIBILITY:
Inclusion Criteria:

* young, healthy volunteers who gave written informed consent - students of health related professions who wear facial mask for at least six hours a day durnig their internship/practice in health care institutions

Exclusion Criteria:

* skin disease, skin damage on measurement sites
* use of corticosteroids, antihistamines and immunomodulators a month prior the inclusion and during the trial
* use of emollients three days prior the inclusion in the trial
* non-adherence to the trial protocol
* exposure to artificial and excessive natural UV radiation
* pregnancy and lactation
* skin cancer
* immunosuppression

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy students of health related professions who wear facial mask daily for at least six hours durnig their internship/practice in health care institutions.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Transepidermal water loss change | Weekly measurements for the duration of six weeks
  Tewameter will be used to assess skin barrier function as a measurement of the water loss (g/hm2).
Stratum corneum hydration change | Weekly measurements for the duration of six weeks
  Corneometer will be used to estimate skin dryness. It is a relative measurement and uses arbitrary units (AU).
Skin erythema change | Weekly measurements for the duration of six weeks
  Mexameter will be used to assess erythema. It is a relative measurement and uses arbitrary units (AU).
Melanin content change | Weekly measurements for the duration of six weeks
  Mexameter will be used to assess skin melanin content. It is a relative measurement and uses arbitrary units (AU).
Participants' reported facial skin changes | Weekly measurements for the duration of six weeks
  Structured interview to determine if participants developed adverse events related to mask wearing (such as dryness, erythema, rash, scaling, pruritus, pain/burning, changes in texture or colour, ulcers etc.) between two measurement time-points.
Sebum level changes | Weekly measurements for the duration of six weeks
  Sebumeter will be used to assess sebum levels. It is a relative measurement and uses arbitrary units (AU).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Montero-Vilchez T, Cuenca-Barrales C, Martinez-Lopez A, Molina-Leyva A, Arias-Santiago S. Skin adverse events related to personal protective equipment: a systematic review and meta-analysis. J Eur Acad Dermatol Venereol. 2021 Oct;35(10):1994-2006. doi: 10.1111/jdv.17436. Epub 2021 Jun 29. PMID 34077565
- [Background] Park SR, Han J, Yeon YM, Kang NY, Kim E. Effect of face mask on skin characteristics changes during the COVID-19 pandemic. Skin Res Technol. 2021 Jul;27(4):554-559. doi: 10.1111/srt.12983. Epub 2020 Nov 20. PMID 33217053
- [Background] Elston DM. Occupational skin disease among health care workers during the coronavirus (COVID-19) epidemic. J Am Acad Dermatol. 2020 May;82(5):1085-1086. doi: 10.1016/j.jaad.2020.03.012. Epub 2020 Mar 18. No abstract available. PMID 32171807
- [Background] Akl J, El-Kehdy J, Salloum A, Benedetto A, Karam P. Skin disorders associated with the COVID-19 pandemic: A review. J Cosmet Dermatol. 2021 Oct;20(10):3105-3115. doi: 10.1111/jocd.14266. Epub 2021 Jul 1. PMID 34077629